CLINICAL TRIAL: NCT05029453
Title: A Prospective, Multicenter, Randomized Controlled Study of Apatinib Combined With Chemotherapy Versus Chemotherapy in Second-line Gastric Cancer Receiving Prior Anti-PD-1 Therapy
Brief Title: Apatinib Combined With Chemotherapy Versus Chemotherapy in Second-line Gastric Cancer Receiving Prior Anti-PD-1 Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Tao Zhang, Chief of gastrointestinal oncology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIONEER
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Gastric Cancer; Randomized Controlled Study
Keywords: apatinib; chemotherapy; prior anti-PD-1 therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): apatinib combine with chemotherapy. Apatinib: initial dose: 500mg,oral,once a day, after meal ( try to take the medicine at the same time each day) Recommended chemotherapy: docetaxel(60/75 mg/m2, d1, q3w)、albuminbound paclitaxel(125mg/m2, d1, d8, q3w) or (260mg/m2, d1, q3w)。
  Interventions: Drug: Apatinib
- Control Gtoup (No Intervention): chemotherapy Recommended chemotherapy: docetaxel(60/75 mg/m2, d1, q3w)、albuminbound paclitaxel(125mg/m2, d1, d8, q3w) or (260mg/m2, d1, q3w)。

INTERVENTIONS:
Drug: Apatinib — In experimental group, the drug used with apatinib and chemotherapy.
  Arms: Experimental Group

SUMMARY:
The study is a multicenter, open-label, randomized controlled clinical study. The purpose of the study is to evaluate the efficacy and safety of apatinib combined with chemotherapy versus chemotherapy in second-line gastric cancer receiving prior anti-PD-1 therapy.

DETAILED DESCRIPTION:
60 patients who meet the inclusion criteria will receive apatinib combine with chemotherapy or chemotherapy until the disease progresses or intolerable.

Apatinib: initial dose: 500mg,oral,once a day, after meal (try to take the medicine at the same time each day)

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, Female or Male;
2. Pathologically diagnosed gastric or gastroesophageal junction adenocarcinoma (GEJ).
3. Failure or intolerance of first-line chemotherapy which requires that the first-line chemotherapy regimen include the scheme based on anti-PD-1 drugs for no less than 2 months (Definition of treatment failure: intolerence of toxic side effects; disease progression during treatment; Or recurrence after the end of treatment.) Note: (1)The treatment of each line advanced disease includes one or more drugs with a medication time ≥ 1 cycle. (2) Early adjuvant/neo-adjuvant therapy is allowed. If recurrence occurs during adjuvant/neoadjuvant therapy or within ≤24 weeks after completion, adjuvant/neoadjuvant therapy is considered to be a first-line pre-systemic chemotherapy for advanced disease. (3) Early-stage immunotherapy, combined chemotherapy or combined targeted drugs are allowed (except for VEGFR inhibitors).
4. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria
5. ECOG performance status 0-1.
6. An expected survival of > 12 weeks.
7. Has adequate sufficient organ and bone marrow functions.
8. Patients whose adverse events caused by previous treatment have recovered to <= CTCAE 1 degree; And the interval between receiving nitroso or mitomycin ≥6 weeks; Receiving other cytotoxic drugs, radiotherapy or surgery ≥ 4 weeks, and the wound has healed completely.
9. Fertile female subjects must undergo a serum-negative pregnancy test within 72 hours before starting the study drug
10. Patients have agreed and signed the informed consent. Willingness and able to follow the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

1. It is known that it's allergic to any test drug and its excipients.
2. Previously received anti-angiogenic therapy, such as Ramucirumab and apatinib.
3. patients with uncontrolled large amount of exudate [chest, pericardium, abdominal cavity]
4. Patients with partial or complete gastrointestinal obstruction.
5. Hypertension, which cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg).
6. Patients with uncontrolled clinical symptoms or diseases of the heart.
7. In the first 3 months of the study, patients who had significant clinical bleeding symptoms or had definite bleeding tendency; History of gastrointestinal perforation and/or fistulae within 6 months prior to medications.
8. Long term use of aspirin, clopidogrel and other antiplatelet drugs, or warfarin and other anticoagulants;
9. Received other therapy within 4 weeks.
10. The patients who received systemic treatment with Chinese herbal medicine or immunomodulatory drugs
11. According to the research's judgement, there are patients who seriously endanger the safety of patients or affect the patients who complete.(such as uncontrolled hypertension、diabetes、thyroid disease, etc)
12. The patient has a serious or non healing wound or peptic ulcer or bone fracture;
13. A patient with other malignancies within 3 years.
14. patients whose adverse events (except hair loss) caused by previous treatment have not recovered to <= CTCAE 1 degree;
15. The researchers considered unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-26 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival [PFS] | 36 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
Objective tumor response rate [ORR] | 1year
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
disease control rate [DCR] | 1year
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）
Duration of response [DoR] | 1year
  Duration of response
overall survival [OS] | 3year
  OS is defined as the length of time from random assignment to death or to last contact.
Adverse Events [AEs] | 1year
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Shi Q, de Gramont A, Grothey A, Zalcberg J, Chibaudel B, Schmoll HJ, Seymour MT, Adams R, Saltz L, Goldberg RM, Punt CJ, Douillard JY, Hoff PM, Hecht JR, Hurwitz H, Diaz-Rubio E, Porschen R, Tebbutt NC, Fuchs C, Souglakos J, Falcone A, Tournigand C, Kabbinavar FF, Heinemann V, Van Cutsem E, Bokemeyer C, Buyse M, Sargent DJ. Individual patient data analysis of progression-free survival versus overall survival as a first-line end point for metastatic colorectal cancer in modern randomized trials: findings from the analysis and research in cancers of the digestive system database. J Clin Oncol. 2015 Jan 1;33(1):22-8. doi: 10.1200/JCO.2014.56.5887. Epub 2014 Nov 10. PMID 25385741
- [Background] Salati M, Di Emidio K, Tarantino V, Cascinu S. Second-line treatments: moving towards an opportunity to improve survival in advanced gastric cancer? ESMO Open. 2017 Jul 19;2(3):e000206. doi: 10.1136/esmoopen-2017-000206. eCollection 2017. PMID 29209523
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of gastric adenocarcinoma. Nature. 2014 Sep 11;513(7517):202-9. doi: 10.1038/nature13480. Epub 2014 Jul 23. PMID 25079317
- [Background] Yan Y, Cao S, Liu X, Harrington SM, Bindeman WE, Adjei AA, Jang JS, Jen J, Li Y, Chanana P, Mansfield AS, Park SS, Markovic SN, Dronca RS, Dong H. CX3CR1 identifies PD-1 therapy-responsive CD8+ T cells that withstand chemotherapy during cancer chemoimmunotherapy. JCI Insight. 2018 Apr 19;3(8):e97828. doi: 10.1172/jci.insight.97828. eCollection 2018 Apr 19. PMID 29669928
- [Background] Shiono A, Kaira K, Mouri A, Yamaguchi O, Hashimoto K, Uchida T, Miura Y, Nishihara F, Murayama Y, Kobayashi K, Kagamu H. Improved efficacy of ramucirumab plus docetaxel after nivolumab failure in previously treated non-small cell lung cancer patients. Thorac Cancer. 2019 Apr;10(4):775-781. doi: 10.1111/1759-7714.12998. Epub 2019 Feb 27. PMID 30809973
- [Background] Park SE, Lee SH, Ahn JS, Ahn MJ, Park K, Sun JM. Increased Response Rates to Salvage Chemotherapy Administered after PD-1/PD-L1 Inhibitors in Patients with Non-Small Cell Lung Cancer. J Thorac Oncol. 2018 Jan;13(1):106-111. doi: 10.1016/j.jtho.2017.10.011. Epub 2017 Oct 31. PMID 29101058
- [Background] Schvartsman G, Peng SA, Bis G, Lee JJ, Benveniste MFK, Zhang J, Roarty EB, Lacerda L, Swisher S, Heymach JV, Fossella FV, William WN. Response rates to single-agent chemotherapy after exposure to immune checkpoint inhibitors in advanced non-small cell lung cancer. Lung Cancer. 2017 Oct;112:90-95. doi: 10.1016/j.lungcan.2017.07.034. Epub 2017 Aug 3. PMID 29191606
- [Background] Harada D, Takata K, Mori S, Kozuki T, Takechi Y, Moriki S, Asakura Y, Ohno T, Nogami N. Previous Immune Checkpoint Inhibitor Treatment to Increase the Efficacy of Docetaxel and Ramucirumab Combination Chemotherapy. Anticancer Res. 2019 Sep;39(9):4987-4993. doi: 10.21873/anticanres.13688. PMID 31519605